CLINICAL TRIAL: NCT01834521
Title: Web-based Screening and Tailored Support for Breast Cancer Patients at the Onset of the Survivorship Phase
Brief Title: Web-based Screening and Tailored Support
Acronym: ENCOURAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ENCOURAGE2-2012; NL41408.042.12 (Other: ABR form Medical Ethical Committee)
Record Dates: First submitted 2013-04-09; First posted 2013-04-18 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; psychosocial; website; empowerment
MeSH Terms: conditions — Breast Neoplasms; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based screening and tailored support (Experimental): A personalized website (username/password) will become available to patients assigned to the intervention arm for 12 subsequent weeks. Key features of the website are self-screening, tailored patient education and self-referral. Self-screening will be performed by an online version of the Dutch Distress thermometer (DT) and Problem List (PL). Patients will receive digital feedback on their DT score immediately after test completion together with information regarding problems reported on the PL, (self)help options and possibilities for referral to professional care. Contact information of one of the investigators will also be available to discuss questions, problems and/or referral needs. Patients may also request a telephone call.
  Interventions: Other: Web-based screening and tailored support
- Standard care (No Intervention): Patients assigned to standard convalescent care will receive the usual follow-up care delivered by their treating oncologists. Patients will be referred to psychosocial or allied care by their oncologist and/or oncology nurse if certain physical and/or psychosocial problems require more in-depth professional care

INTERVENTIONS:
Other: Web-based screening and tailored support
  Arms: Web-based screening and tailored support

SUMMARY:
The ever expanding breast cancer survivor population urges the health care system to develop (cost-)effective screening and management of convalescent care needs that can be easily implemented in conventional follow-up care. Internet-delivered systems may be well-equipped to meet these demands. The aim of the current study is to assess the effectiveness of a web-based support system. Key features of this system are patient self-screening of physical and psychosocial problems, tailored patient education on reported problems and self-referral to professional care. In this era of high internet usage, we expect that internet is a highly suitable medium to provide tailored support for breast cancer patients and will empower the patient to take control over their convalescence.

ELIGIBILITY:
Inclusion Criteria:

* Adult female breast cancer patients (aged ≥ 18 years of age).
* Recent completion (≤6 months) of (neo)adjuvant chemotherapy for primary breast cancer
* Ability to comprehend Dutch (both reading and writing).
* Access to internet (e.g. at home, via family or friends)
* Informed consent provided

Exclusion Criteria:

• Chemotherapy treatment with palliative intent or recurrent breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from 6 to 12 weeks follow-up in optimism and control over the future | 6 and 12 weeks
  Patients' optimism and control over the future will be measured by the subscale 'increased optimism and control over the future' of the 'Constructs Empowering Outcomes Questionnaire'. The subscale 'optimism and control over the future' represents a single concept/outcome measure. The concept cannot be assessed at baseline due to the retrospective nature of the questionnaire.

SECONDARY OUTCOMES:
Change from 6 to 12 weeks follow-up in knowledge level | 6 and 12 weeks
  Patient knowledge level will be measured by the subscale 'being better informed' of the 'Constructs Empowering Outcomes Questionnaire'. The concept cannot be assessed at baseline due to the retrospective nature of the questionnaire.
Change from 6 weeks to 12 weeks follow-up in acceptance of problems | 6 and 12 weeks
  Patients' acceptance of their problems will be measured by the subscale 'improved acceptance of the illness' of the 'Constructs Empowering Outcomes Questionnaire'. The concept cannot be assessed at baseline due to the retrospective nature of the questionnaire.
Change from baseline to 12 weeks follow-up in quality of life | Baseline and 12 weeks follow-up
  Cancer-specific quality of life will be measured by the EORTC QLQ-C30 (version 3.0) questionnaire.
Change from baseline to 12 weeks follow-up in psychological distress | Baseline and 12 weeks follow-up
  Psychological distress will be measured by the Dutch Distress Thermometer and Problem List.

CONTACTS AND LOCATIONS:
Overall Officials: A.K.L. Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands